CLINICAL TRIAL: NCT00269035
Title: A Parallel Study to Investigate Dopaminergic D2 and Serotoninergic 5HT2A Receptor Occupancy at Stable Plasma Concentrations of SB-773812 After Repeated Doses in Schizophrenic Patients. Relationship With Pharmacokinetics and Efficacy Readouts.
Brief Title: SPECT Study With SB-773812 In Schizophrenic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 773812/007
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
Keywords: SB-773812; SPECT; D2 RO; pharmacokinetics; schizophrenic patients; 5HT2A RO
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Experimental): Subjects in group 1 will receive SB-773812 tablet once daily till still steady Cp
  Interventions: Drug: SB773812
- Treatment Group 2 (Experimental): Subjects in group 2 will receive SB-773812 tablets once daily over 6 weeks. Risperidone tablets 6 mg once daily from Days 1-7 two tablets of 3 mg and days 8 until stable Cp 6 mg tablets
  Interventions: Drug: SB773812; Drug: Risperidone

INTERVENTIONS:
Drug: SB773812 — SB-773812 tablets will be available with dose strength of 60 mg
Drug: Risperidone — Risperidone tablets will be available with dose strength of 3 and 6 mg
  Arms: Treatment Group 2

SUMMARY:
This study is being conducted in 2 groups of schizophrenic patients: in group 1 the relationship between the dopaminergic D2 receptor occupancy (D2 RO ) and serotoninergic 5HT2A receptor occupancy at stable plasma concentration (Cp) of SB-773812 will be investigated using SPECT scan in up to 15 chronic schizophrenic patients in an open- label design. In group 2 up to 80 patients will receive SB-773812 or Risperidone for 6 weeks to obtain at least 10 patients showing clinical improvement with SB-773812. The relationship of D2 RO, measured at steady state after chronic dosing at Cmax (6+/-2 h) and Ctrough (24+/-4 h), and PK at steady state after repeated doses, to efficacy readouts will be investigated. The SB-773812 dose administered will be selected as the highest dose proven to be safe and well tolerated from a previous study.

ELIGIBILITY:
Inclusion criteria:

* schizophrenic patients as diagnosed by DSM IV criteria.
* In group 2, subject has schizophrenia or schizophreniform disorder and show moderate disease exacerbation, a PANSS score > 65 and a score in the PANSS positive scale (PANSS-P) =25.
* Women of childbearing potential must agree to acceptable method of birth control.

Exclusion criteria:

* Subject shows severe exacerbation, extreme instability, high risk for suicide or serious violent behaviour.
* Any clinically or laboratory significant abnormality.
* Subjects receiving a radiation dose from other activities of more than 10 mSv over any 3 year period.
* Subjects with organic brain disease and history of severe head trauma.
* Heart pacemaker, metallic prosthesis or other metallic body implants.
* Significant head deformity.
* Smokers with associated COPD.
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease.
* History of cholecystectomy or biliary tract disease.
* Positive for HBV, HCV or HIV.
* Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2005-06-21 (Actual); Primary Completion 2007-05-26 (Actual); Study Completion 2007-05-26 (Actual)

PRIMARY OUTCOMES:
To investigate in schizophrenic patients the relationship between D2 RO, 5HT2A RO and stable plasma concentrations of SB-773812 (gr.1) and the relationship of D2 RO and PK over time at steady state to efficacy readouts after 6 w treatment (gr.2) | 6 weeks

SECONDARY OUTCOMES:
To assess the effect of 6 week treatment of SB-773812 on clinical symptoms as measured by Positive and Negative Symptoms Scale (PANSS), cognitive performance and CGI Severity and Improvement as a function of duration of dosing (group 2). | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Mataro (Barcelona)
  - GSK Investigational Site, Sant Boi de Llobregat
  - GSK Investigational Site, Vic (Barcelona)

REFERENCES:
- See also: Results for study 773812/007 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/773812/007?search=study&search_terms=773812%2F007#rs